CLINICAL TRIAL: NCT02464215
Title: Comparison of the Laparoscopy-Assisted Distal Gastrectomy(LADG) and Open Distal Gastrectomy(ODG) for Locally Advanced Gastric Cancer
Brief Title: Effect of Laparoscopy-Assisted Distal Gastrectomy for Locally Advanced Gastric Cancer
Acronym: SWEET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Beijing Friendship Hospital (Other); Beijing Shijitan Hospital, Capital Medical University (Other); Xuanwu Hospital, Beijing (Other); Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, Xiangqian Su, Principal Investigator, Peking University Cancer Hospital & Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XM201309
Record Dates: First submitted 2015-06-01; First posted 2015-06-08 (Estimated); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; D2; laparoscopic; open; surgery
MeSH Terms: conditions — Stomach Neoplasms | interventions — Conversion to Open Surgery; Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- open surgery (Active Comparator): Conventional procedure,Open surgery
  Interventions: Procedure: open surgery
- laparoscopic surgery (Experimental): Minimum invasive procedure，Laparoscopic surgery
  Interventions: Procedure: laparoscopic surgery

INTERVENTIONS:
Procedure: open surgery — Subtotal gastectomy (dissect more than 2/3 of stomach and total omentectomy) and D2 lymph node dessection(around common hepatic artery, celiac artery, proximal part of splenic artery, hepatoduodenal ligament, superior mesenteric vein) will be performed basically.
  Other Names: ODG
  Arms: open surgery
Procedure: laparoscopic surgery — Patients in this arm undergo radical resection of gastric cancer in laparoscopic surgery.10 mm trocar under umbilicus, 12 mm and 5 mm trocar at the right flank area are inserted into abdominal wall. Another two 5 mm trocar are inserted into the both midline of subcostal line. The devices for operation are inserted through the trocars. Subtotal gastrectomy (dissect more than 2/3 of stomach and total omentectomy) and D2 lymph node dissection (around common hepatic artery, celiac artery, proximal part of splenic artery, hepatoduodenal ligament, superior mesenteric vein) will be performed basically. Dissected stomach and lymph node are collected through additional 5-10 cm incision at the preexisting epigastric incision.
  Other Names: LADG
  Arms: laparoscopic surgery

SUMMARY:
The purpose of this study is to evaluate the effect and safety of laparoscopy-assisted D2 radical surgery for distal advanced gastric cancer.

DETAILED DESCRIPTION:
In both arms,subtotal gastrectomy (dissect more than 2/3 of stomach and total omentectomy) and D2 lymph node dissection (around common hepatic artery, celiac artery, proximal part of splenic artery (4d, 4sb), hepatoduodenal ligament, superior mesenteric vein) wiil be performed basically. As a general rule, Billroth I or BillrothII methods will be used for gastric reconstruction for all cases. For anastomosis, absorbable suture is used. Anastomotic diameter is 5~6 cm length. Drainage tube is inserted through the right flank area and additional drainage tubes can be inserted as needed.

ELIGIBILITY:
Inclusion Criteria:

1. Age: older than 18 years old，including 18 years old
2. Pathologic finding by gastric endoscopy: confirmed gastric adenocarcinoma (papillary adenocarcinoma, tubular adenocarcinoma, mucinous adenocarcinoma, signet ring cell carcinoma, poorly differentiated adenocarcinoma)
3. Cancer core: located at lower part of stomach
4. Preoperative cancer stage : cT2-4a,N0-3,M0 (according to AJCC-7th TNM staging)
5. surgery：subtotal gastrectomy (dissect more than 2/3 of stomach and total omentectomy) and D2 lymph node dissection
6. ASA score: ≤ 3;ECOG performance status 0/1
7. Informed consent patients (explanation about our clinical trials is provided to the patients or patrons, if patient is not available)

Exclusion Criteria:

1. Concurrent cancer patients or patient who was treated due to other types of cancer before the patient was diagnosed as a gastric cancer patient
2. Patient who was treated by other types of treatment methods, such as chemotherapy, immunotherapy, or radiotherapy
3. Patient who was received upper abdominal surgery (except, laparoscopic cholecystectomy)
4. Patient who was treated because of systemic inflammatory disease
5. Pregnant patient or lactating women
6. Patient who suffer from bleeding tendency disease, such as hemophilia or patient taking anti-coagulant medication due to deep vein thrombosis
7. serious mental illness
8. gastric surgery (including for gastric ESD / EMR)
9. imaging examinations showed regional integration lymph nodes (maximum diameter ≥ 3cm)
10. other malignant diseases in 5 years
11. have unstable angina or myocardial infarction within six months
12. have cerebral infarction or cerebral hemorrhage within 6 months
13. sustained systemic glucocorticoid treatment history within 1 month
14. have other diseases needed operative treatment at the same time
15. complications (bleeding, perforation, obstruction) required emergency surgery
16. Pulmonary function tests FEV1 <50% of predicted value.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2014-03-01; Primary Completion 2020-08-31 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative complication rate | 30 days
  Surgical complications within 30 days after surgery

SECONDARY OUTCOMES:
3-year disease free survival rate | 3 years
  3-year disease free survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Xiangqian Su, professor, Principal Investigator — Department of Minimally Invasive Gastrointestinal Surgery, Peking University Cancer Hospital & Institute
Locations (1):
- Department of Minimally Invasive Gastrointestinal Surgery, Peking University Cancer Hospital & Institute, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Xing J, Cai J, Wang X, Zhang N, An D, Li F, Cui M, Niu L, Gao C, Fan Q, Ren S, Zhang Z, Su X; SWEET trial group. Long-term outcomes of laparoscopic versus open distal gastrectomy for patients with advanced gastric cancer in North China: a multicenter randomized controlled trial. Surg Endosc. 2024 Sep;38(9):4976-4985. doi: 10.1007/s00464-024-10952-2. Epub 2024 Jul 9. PMID 38981881
- [Derived] Wang Z, Xing J, Cai J, Zhang Z, Li F, Zhang N, Wu J, Cui M, Liu Y, Chen L, Yang H, Zheng Z, Wang X, Gao C, Wang Z, Fan Q, Zhu Y, Ren S, Zhang C, Liu M, Ji J, Su X. Short-term surgical outcomes of laparoscopy-assisted versus open D2 distal gastrectomy for locally advanced gastric cancer in North China: a multicenter randomized controlled trial. Surg Endosc. 2019 Jan;33(1):33-45. doi: 10.1007/s00464-018-6391-x. Epub 2018 Nov 1. PMID 30386984